CLINICAL TRIAL: NCT06080724
Title: Efficacy of Intralesional Bleomycin Alone and in Combination With Dexamethasone in Infantile Haemangiomas
Acronym: hemangioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Muhammad Sharif, PROFESSOR, King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2023-09-09; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Comparison of Efficacy of Sclerotherapy in Infantile Hemangioma
Keywords: infantile hemangioma; Bleomycin; Sclerotherapy; Dexamethasone; Combined sclerotherapy
MeSH Terms: conditions — Hemangioma, Capillary

STUDY DESIGN:
Intervention Model Description: A randomized control trial study was conducted on patients of haemangiomas of pediatric age group coming to pediatric surgery ward, KEMU/Mayo hospital, Lahore. Patients were randomized in two study groups A and B. The Lottery method was used for allocation of patients where the patient was given allocated treatment regimen after opening the sealed envelope. Each group contained 57 of patients. Patients in the group A were given intralesional bleomycin combined with dexamethasone and in the group B intralesional bleomycin alone after taking aseptic and antiseptic measures. T
Who Masked: Participant, Outcomes Assessor
Masking Description: participants were up to age of 12 years so they automatically got masked. outcome assessors were the teams of doctor working in outpatient department were also masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A with intralesional injection of bleomycin with dexamethasone (Other): Patients in the group A(n=57) were given intralesional bleomycin combined with dexamethasone and The intralesional dose of bleomycin was 1 mg/kg/dose but for haemangiomas on neck and face it was used as 0.5 mg/kg/dose and similarly intralesional dexamethasone was given as 0.8-1.6 mg/kg/dose. The Length, Width, Height and volume of haemangioma was measured in centimeters using a vernier calliper. The decrease in size was graded from 1-5 where 1=<50% decrease, 2=50-75%, 3=75-90%, 4=>90% but <100% and 5= 100% resolution. The data collection sheet included patent's age, sex, length, width, height, volume, site of haemangioma, dose of bleomycin, dexamethasone, clinical response being efficacious or non-efficacious as per operational definition and time taken to resolve for each patient.
  Interventions: Drug: Comparison of intralesional injection of bleomycin alone and combined with injection dexamethasone
- Group B WITH INTRALESIONAL INJECTION OF BLEOMYCIN (Other): Patients in the group B(n=57) intralesional bleomycin alone after taking aseptic and antiseptic measuresThe intralesional dose of bleomycin was 1 mg/kg/dose but for haemangiomas on neck and face it was used as 0.5 mg/kg/dose.The Length, Width, Height and volume of haemangioma was measured in centimeters using a vernier calliper. The decrease in size was graded from 1-5 where 1=<50% decrease, 2=50-75%, 3=75-90%, 4=>90% but <100% and 5= 100% resolution. The data collection sheet included patent's age, sex, length, width, height, volume, site of haemangioma, dose of bleomycin, dexamethasone, clinical response being efficacious or non-efficacious as per operational definition and time taken to resolve for each patient.
  Interventions: Drug: Comparison of intralesional injection of bleomycin alone and combined with injection dexamethasone

INTERVENTIONS:
Drug: Comparison of intralesional injection of bleomycin alone and combined with injection dexamethasone — already described

SUMMARY:
Objective:

This study is intended to compare the outcome of intralesional bleomycin with dexamethasone versus the bleomycin alone in infantile haemangioma.

Materials and Methods:

This RCT was performed after the ethical approval at the pediatric surgery department of KEMU/Mayo hospital Lahore. 114 patients were enrolled in two groups A and B. Both groups contained 57 patients each. Group A was administered intralesional bleomycin with dexamethasone and group B was given intralesional bleomycin alone with a space of 4 weeks. Selection of patients was made according to inclusions and exclusion criteria.

DETAILED DESCRIPTION:
Introduction:

Infantile haemangioma (IH) is a common tumor found in children. The history of this tumor consists of an early phase of growth followed by slow resolution over a period of three to seven years but can extend up to 12 years. Therapeutic intervention is usually not required in infantile hemangiomas due to spontaneous regression. In about 10 to 15% of cases IH located in the perineal, airway or periocular areas, or hemangiomas associated with complications of ulceration, intervention is necessary. Another reason for intervention in these hemangiomas is the probability of scar formation with complete or incomplete spontaneous involution. Currently available treatment options for IH range from topical, intralesional, systemic and laser therapies to surgery based on the stage and presentation of the tumor. The choice of treatment must be carefully selected after comparing the merits and risks of each modality through a patient-specific approach.

OPERATIONAL DEFINITION:

Infantile Haemangioma: is a benign vascular proliferative disorder which has an early period of proliferation and then regresses spontaneously. They are found during the infancy and are considered medically benign lesions.

Efficacy: The desired effect obtained after giving a treatment is termed as efficacy. Efficacy of the treatment was measured in terms of reduction of the size of haemangioma which in turn was assessed by measuring length, width, height and volume every month to a period of one year. The decrease in size was graded on 5 point scale where 1= < 50% reduction, 2= 50-75%, 3= 75-90%, 4= >90% but < 100% and 5= 100%[17]. The complete flattening of haemangioma was considered as resolution of the lesion and at least the reduction in size of grade 2 results was labelled as the treatment being efficacious.

Intralesional Injection: After aseptic measures the injection was administered using a 26 gauge needle by directly injecting into the haemangioma in 4 different directions (the lesion was divided into 4 imaginary quadrants by drawing to perpendicular lines) through the single puncture point. Sterile gauze was used for pressure until the bleeding stopped.

Dosage: The intralesional dose of bleomycin was 1 mg/kg/dose but for haemangiomas on neck and face it was used as 0.5 mg/kg/dose and similarly intralesional dexamethasone was given as 0.8-1.6 mg/kg/dose. Both the drugs were administered intralesionally every 4 weeks. Every patient was checked for sensitivity to the drugs.

Treatment Response: The response of the treatment was evaluated by measuring Length, Width, Height and Volume. The length, width and height was measured using a vernier calliper in centimeters before administering the first injection and then after every 4 weeks following each injection.

Hypothesis:

The intralesional bleomycin combined with dexamethasone is more efficacious than intralesional bleomycin alone in infantile haemangioma.

Material and Methods:

Study Design: It was be a Randomized Controlled Trial.

Study Setting: The study was conducted in Pediatric surgery department, KEMU/Mayo Hospital Lahore.

Duration Of The Study: 1 year after the approval of the synopsis. Sampling Technique: Probability simple random sampling. Sample Size: Sample size of 114 patients ( 57 patients in each group ) is estimated by using 95% confidence level, 10% absolute precision with expected percentage of intralesional bleomycin combined with dexamethasone as 100%[15] and intralesional bleomycin alone as 82%[10] .

n = Z1-α/2 [ P1 (1- P1) + P2 (1- P2) ] d2 Where n = sample size P1 = population proportion I = 100% P2 = population proportion II = 82% Z1-α/2 = confidence level 95% = 1.96 d = absolute precision 10%

Sample Selection:

Inclusion Criteria:

1. Patients with haemangiomas presenting to pediatric surgery department KEMU/Mayo hospital Lahore with size equal or more than 1 cm.
2. Patients </= 12 years and above 1 month of age.

Exclusion Criteria:

1. Patients who had undergone any surgical procedure for haemangiomas proved from the history.
2. Patients with chronic respiratory conditions confirmed by history, symptoms and physical examination.
3. The diagnosed case of pulmonary fibrosis.
4. Patients sensitive to bleomycin proved upon giving a test dose.

DATA COLLECTION PROCEDURE:

Permission was taken from the ethical review board. Patients were selected as per inclusion and exclusion criteria. Written informed consent was taken from parents/guardians regarding inclusion in study and sharing of data after counseling about the procedure, drug effects and follow up. A randomized control trial study was conducted on patients of haemangiomas of pediatric age group coming to pediatric surgery ward, KEMU/Mayo hospital, Lahore. Patients were randomized in two study groups A and B. The Lottery method was used for allocation of patients where the patient was given allocated treatment regimen after opening the sealed envelope. Each group contained 57 of patients. Patients in the group A were given intralesional bleomycin combined with dexamethasone and in the group B intralesional bleomycin alone after taking aseptic and antiseptic measures. The intralesional dose of bleomycin was 1 mg/kg/dose but for haemangiomas on neck and face it was used as 0.5 mg/kg/dose and similarly intralesional dexamethasone was given as 0.8-1.6 mg/kg/dose. The Length, Width, Height and volume of haemangioma was measured in centimeters using a vernier calliper. The decrease in size was graded from 1-5 where 1=<50% decrease, 2=50-75%, 3=75-90%, 4=>90% but <100% and 5= 100% resolution. The data collection sheet included patent's age, sex, length, width, height, volume, site of haemangioma, dose of bleomycin, dexamethasone, clinical response being efficacious or non-efficacious as per operational definition and time taken to resolve for each patient.

DATA ANALYSIS PROCEDURE:

Data was entered and processed by using SPSS-26. Quantitative variable like age, length, width, height, volume, grades of improvement and time for resolution was presented as mean+SD . Qualitative variables like site of haemangioma, gender and efficacy was described using frequencies and percentages. Comparison of two groups "intralesional bleomycin alone" and "intralesional bleomycin combined with dexamethasone" was done by applying independent sample t-test. P-value if <0.05 was taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haemangioma with size equal or more than 1 c
* Less than 12 years and above 1 month of age.

Exclusion Criteria:

* Patients with previous surgical procedure for haemangiomas
* Patients with chronic respiratory conditions confirmed by history, symptoms and physical examination.
* The diagnosed case of pulmonary fibrosis.
* Patients sensitive to bleomycin proved upon giving a test dose

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Decrease in size of lesion | 1 year
  The Length, Width, Height and volume of haemangioma was measured in centimeters using a vernier calliper. The decrease in size was graded from 1-5 where 1=<50% decrease, 2=50-75%, 3=75-90%, 4=>90% but <100% and 5= 100% resolution.

CONTACTS AND LOCATIONS:
Locations (1):
- department of pediatric surgery King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided